CLINICAL TRIAL: NCT05523531
Title: Description of Symptoms, Impact on Quality of Life, Ophthalmological Examination and Treatment of Patients With Neuropathic Eye Pain Associated With Dry Eye: a Prospective Single-center Long-term Follow-up Study of a Series of Cases Previously Included in the QUALVIDON Study
Brief Title: Prospective Single-center Long-term Follow-up Study of a Series of Cases Previously Included in the QUALVIDON Study
Acronym: QUALVIDON2
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SDN_2022_7
Record Dates: First submitted 2022-08-08; First posted 2022-08-31 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Dry Eye; Neuropathic Pain
Keywords: Dry eye; Neuropathic eye pain; Quality of Life
MeSH Terms: conditions — Dry Eye Syndromes; Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with characteristics of idiopathic neuropathic eye pain associated with dry eye: Previously included in the QUALVIDON study
  Interventions: Other: Self-administered questionnaires; Procedure: Bilateral ophthalmologic examination

INTERVENTIONS:
Other: Self-administered questionnaires — * Neuropathic Eye Pain Questionnaire
  * 5-item Dry Eye Evaluation Questionnaire (DEQ-5)
  * Visual Impact Assessment Questionnaire
  * Concise Ophthalmic Pain Questionnaire
  * Questionnaire to evaluate the effectiveness and tolerance of treatments
  * Chronic pain questionnaire
Procedure: Bilateral ophthalmologic examination — * Examination of the ocular surface and eyelids Slit lamp with fluorescein instillation: Oxford scheme and Break-up time, Schirmer's test, Oxybuprocaine test
  * Lipiview® test
  * Examination of corneal sensitivity with the Cochet-Bonnet esthesiometer
  * In vivo morphological examination of the subepithelial nerve plexus of the cornea by confocal microscopy

SUMMARY:
Dry eye affects millions of people around the world. Some dry eye patients complain of neuropathic eye pain that can affect their quality of life.

From August 2016 to June 2017, the QUALVIDON study (NCT03296111), conducted at the Adolphe de Rothschild Foundation Hospital, assessed pain and its impact on quality of life using self-administered questionnaires in a series of dry eye patients. This 2nd study, entitled QUALVIDON2, focuses on the outcome of patients previously included in QUALVIDON.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously included in the QUALVIDON study with the following characteristics:
* With characteristics of idiopathic neuropathic eye pain associated with dry eye
* Give informed consent
* Affiliated or beneficiary of the french social security

Exclusion Criteria:

* Pregnant or nursing woman
* Patient under legal protection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients previously included in the QUALVIDON study, with characteristics of idiopathic neuropathic eye pain associated with dry eye
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Assessment of neuropathic eye pain | at 5 years follow-up
  Total score of the french neuropathic eye pain questionnaire (QDON) Range from 0 to 28. A score with higher value reflects a more severe disease.

SECONDARY OUTCOMES:
Assessment of Oxford score | at 5 years follow-up
  Oxford score (range from 0 to V). Interpretation: 0= mild symptoms to V= severe symptoms.
Assessment of Schirmer's test | at 5 years follow-up
  Schirmer's test (in millimeters)
Assessment of Tear break up time | at 5 years follow-up
  Tear break up time (in seconds)
Diagnosis of blepharitis | at 5 years follow-up
  Diagnosis of blepharitis (none or yes: minimal/moderate/severe)
Assessment of Meibomian gland dysfunction | at 5 years follow-up
  Meibomian gland dysfunction (none or yes: minimal/ moderate/severe)
Assessment of the thickness of tear film lipid Layer | at 5 years follow-up
  Characterization of the thickness of the tear film lipid Layer (evaluated by Lipiview® and quantified by the device in nm)
Diagnosis of atrophy of the Meibomian glands | at 5 years follow-up
  Diagnosis of atrophy of the Meibomian glands (evaluated by Lipiview® and rated by the device, from 0 to 4)
Assessment of corneal sensitivity | at 5 years follow-up
  Corneal sensitivity will be assessed by the Cochet-Bonnet aesthesiometer (in millimeters)
Assessment of dry eye severity | at 5 years follow-up
  Total score of the french version of the DEQ-5 (Dry Eye Questionnaire). Range from 0 to 22. A score with higher value reflects a more severe dryness.
Visual impact of dry eye | at 5 years follow-up
  Total score of the french version of the OSDI (Ocular Surface Disease Index). Range from 0 to 48. A score with higher value reflects a more severe visual impact.
General impact of eye pain | at 5 years follow-up
  Total score of the french version of the modified BPI (Brief Pain Inventory) for ophtalmology.
  Range from 0 to 110. A score with higher value reflects a more severe general impact of the pain.
Psychologic impact of eye pain | at 5 years follow-up
  Total sub-scores of Anxiety (A) and depression (D) of the french version of the HAD (Hospital Anxiety and Depression Scale).
  Scores A (Anxiety): range from 0 to 21. Interpretation: < or = 7: no symptom of anxiety, 8 to 10: uncertain symptomatology, > or = 7: symptoms of anxiety Scores D (Depression): range from 0 to 21. Interpretation: < or = 7: no symptom of depression, 8 to 10: uncertain symptomatology, > or = 7: symptoms of depression
Drug effectivness (pain relief) | at 5 years follow-up
  Pain relief will be assess with a likert type scale (range from 0 = "none" to 5 = "total relief") for each drug
Drug safety | at 5 years follow-up
  Drug safety will be assess with a likert type scale (range from 0 = "none" to 5 = "total safety") for each drug

CONTACTS AND LOCATIONS:
Overall Officials: Serge DOAN, MD, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France